CLINICAL TRIAL: NCT00693485
Title: Safety and Effects of Brimonidine Intravitreal Implant in Patients With Glaucomatous Optic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190342-030D
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Results first posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-03

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Brimonidine Tartrate; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 400 ug Brimonidine Implant (Experimental): 400 ug Brimonidine Tartrate Posterior Segment Drug Delivery system; Applicator System at Day 1 in study eye.
  Interventions: Drug: 400 ug Brimonidine Implant
- 200 ug Brimonidine Implant (Experimental): 200 ug Brimonidine Tartrate Posterior Segment Drug Delivery system; Applicator System at Day 1 in study eye.
  Interventions: Drug: 200 ug Brimonidine Implant
- Sham (no implant) (Sham Comparator): Sham Posterior Segment Drug Delivery system; Applicator System at Day 1 in study eye.
  Interventions: Drug: Sham (no implant)

INTERVENTIONS:
Drug: 400 ug Brimonidine Implant — 400 ug Brimonidine Tartrate Posterior Segment Drug Delivery system; Applicator System at Day 1 in study eye.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 400 ug Brimonidine Implant
Drug: 200 ug Brimonidine Implant — 200 ug Brimonidine Tartrate Posterior Segment Drug Delivery system; Applicator System at Day 1 in study eye.
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 200 ug Brimonidine Implant
Drug: Sham (no implant) — Sham Posterior Segment Drug Delivery system; Applicator System at Day 1 in study eye.
  Arms: Sham (no implant)

SUMMARY:
A multicenter, randomized, patient-masked, sham-controlled evaluation of the safety and effects on visual function of brimonidine intravitreal implant in patients with glaucomatous optic neuropathy. Patients will be followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle glaucoma in one eye
* Visual acuity 20/80 or better
* Intraocular pressure in the study eye ≤ 24 mm Hg
* Glaucomatous visual field loss - 7 dB to - 25 dB

Exclusion Criteria:

* Known allergy to brimonidine tartrate
* Uncontrolled systemic disease or infection of the eye
* Recent eye surgery or injections in the eye
* Female patients who are pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-09; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Artesia, California, United States
- Tel Aviv, Israel

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Started | 25 | 21 | 24
Completed | 25 | 19 | 24
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant) | Total
Number analyzed (Participants) | 25 | 21 | 24 | 70
Age, Customized [Number; unit: Participants]
  <45 years | 0 | 0 | 1 | 1
  Between 45 and 65 years | 9 | 11 | 12 | 32
  >65 years | 16 | 10 | 11 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 10 | 34
  Male | 13 | 9 | 14 | 36
Mean Deviation from Normal Visual Field Using the HFA 24-2 [Mean (Full Range); unit: Decibels (db)] — Mean deviation is the difference between the expected normal visual field compared to the patient's visual field.
  Decibels (db) | -15.5 (5.26) [-28.2 to -6.4] | -14.6 (3.67) [-24.3 to -10.1] | -17.9 (5.09) [-30.9 to -9.4] | -16.0 [-30.9 to -6.4]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With a Visual Field Improvement in the Study Eye
Description: Visual field improvement in the study eye is determined using the Humphrey Field Analyzer (HFA 24-2) full threshold test and clinical expertise. The Humphrey Field Analyzer is a machine that helps to map the field (peripheral) of vision. An improvement is an increase in the field of vision. The percentage of patients with a visual field improvement in the study eye is reported.
Time Frame: Baseline, Month 6
Population: Safety Population: all patients who received 1 dose of study medication or sham treatment
Measure: Number; unit: Percentage of Patients
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Number analyzed (Participants) | 25 | 21 | 24
Percentage of Patients | 12.0 | 9.5 | 4.2

2. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A positive change from baseline indicates an improvement and a negative change from baseline indicates a worsening.
Time Frame: Baseline, Month 6
Population: Safety Population: all patients who received 1 dose of study medication or sham treatment
Measure: Mean (Standard Deviation); unit: Number of Letters Read Correctly
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Number analyzed (Participants) | 25 | 21 | 24
Number of Letters Read Correctly
  Baseline | 76.0 (7.82) | 80.6 (6.20) | 77.3 (7.71)
  Change from Baseline at Month 6 | 2.8 (3.68) | -2.2 (18.35) | 0.3 (5.18)

ADVERSE EVENTS:
Description: For Ocular Adverse Events (AEs), only those in the study eye are reported in the "Other Adverse Events" section. For Serious Adverse Events (SAEs), all ocular events were reported in the SAE section, regardless of the eye.
Arm/Group | 400 ug Brimonidine Implant | 200 ug Brimonidine Implant | Sham (no Implant)
Serious Adverse Events (participants affected / at risk) | 3/25 | 5/21 | 1/24
Other Adverse Events (participants affected / at risk) | 18/25 | 19/21 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 ug Brimonidine Implant (N=25) | 200 ug Brimonidine Implant (N=21) | Sham (no Implant) (N=24)
Arteriospasm coronary (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 400 ug Brimonidine Implant (N=25) | 200 ug Brimonidine Implant (N=21) | Sham (no Implant) (N=24)
Conjunctival haemorrhage (Eye disorders) | 6 | 2 | 3
Intraocular pressure increased (Investigations) | 3 | 2 | 2
Punctate keratitis (Eye disorders) | 4 | 2 | 1
Headache (Nervous system disorders) | 4 | 1 | 0
Conjunctival Hyperaemia (Eye disorders) | 3 | 3 | 3
Hypertension (Vascular disorders) | 3 | 2 | 0
Eye Irritation (Eye disorders) | 3 | 0 | 2
Eye Pain (Eye disorders) | 3 | 1 | 0
Blepharitis (Eye disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 3
Lacrimation Increased (Eye disorders) | 1 | 1 | 2
Conjunctivitis (Eye disorders) | 1 | 2 | 1
Foreign Body Sensation in Eyes (Eye disorders) | 1 | 2 | 0
Vitreous Detachment (Eye disorders) | 0 | 1 | 2
Cataract (Eye disorders) | 0 | 1 | 3
Retinal Pigmentation (Eye disorders) | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.